CLINICAL TRIAL: NCT04059159
Title: Evaluation of the Safety and Clinical Performance of the Gen 2 Connected Catheter - Wireless Urinary Prosthesis for Management of Chronic Urinary Retention
Brief Title: Connected Catheter - Safety and Effectiveness Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigation of this device has been transitioned into a new study by the sponsor. The data generated in this study will not be used to support a marketing application
Sponsor: Spinal Singularity (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIP-0002 (formerly ES-NIH-01)
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Neurogenic Bladder; Urinary Retention; Urologic Diseases
Keywords: catheter; Spinal Cord Injury (SCI)
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Retention; Urologic Diseases; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Connected Catheter Users (Experimental)
  Interventions: Device: Connected Catheter

INTERVENTIONS:
Device: Connected Catheter — Patients will use the Connected Catheter to empty the bladder during the course of treatment.

SUMMARY:
The Connected Catheter is a fully internal, urethral indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization. It is a sterile, extended-use device that resides fully internally to the male lower urinary tract for an intended use life of up to 7 days per catheter.

DETAILED DESCRIPTION:
Spinal Singularity has developed the Connected Catheter System to address several drawbacks of urinary catheters. The Connected Catheter is fully internal, indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization. Each subject will use the Connected Catheter for up to 35-40 days. This includes five device exchange appointments. The appointments are spaced 7 days apart and at each appointment the catheter will be replaced with a new one. Additionally, weekly follow-up will occur for 14 days following the final appointment after the subject discontinues use of study device and reverts to his original catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Males age ≥ 18 with clinical diagnosis of significant urinary retention
2. Must be clinically suitable and capable of safely managing bladder using an intermittent voiding or indwelling strategy

   1. Must have stable urinary management history as determined by the investigator OR:
   2. Must have urodynamic profile suitable for Gen 2 Connected Catheter (including bladder capacity > 200mL without uninhibited bladder contractions)
3. Subject's lower urinary tract anatomy must fall within the ranges serviceable by the Gen 2 Connected Catheter device, as specified in the Investigational Device Instructions for Use (IFU).

Exclusion Criteria:

1. Active symptomatic urinary tract infection, as defined in this clinical investigation protocol (subjects may receive the device after UTI has been treated)
2. Significant risk profile or recent history of urethral stricture (e.g. stricture within past 90 days)
3. Significant risk profile or recent history of clinically significant (uncontrolled) autonomic dysreflexia
4. Significant intermittent urinary incontinence (between catheterizations)
5. Uninhibited bladder contractions and/or Vesicoureteral reflux that is not reliably controlled with medication or alternate therapy (e.g. Botox injection)
6. Pre-existing urinary pathologies and/or morphological abnormalities of the lower urinary tract or bladder (assessed during in-depth medical screening, including cystoscopy and urine analysis)

   1. Urinary tract inflammation or neoplasm
   2. Urinary fistula
   3. Bladder diverticulum (outpouching) > 5cm in size
   4. Chronic pyelonephritis (secondary to upper urinary tract infection(s) within past 6 months)
   5. Impaired kidney function or renal failure
   6. Active gross hematuria
   7. Active urethritis
7. Dependence on an electro-magnetic medical implant (e.g. cardiac pacemaker or implanted drug pump) or external device
8. Any unsuitable comorbidities as determined by the Investigator or complications related to use of certain medications
9. Any physical or cognitive impairments that diminish the subject's ability to follow directions or otherwise safely use the Gen 2 Connected Catheter System
10. Catheter Assessment Tool screening yields unacceptable results

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Device is currently only designed for use by males.
Enrollment: 8 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rancho Los Amigos Rehabiliation Hospital, Downey, California
  - UC San Diego, San Diego, California
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Connected Catheter Users
Started | 8
Completed | 3
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Connected Catheter Users
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White or Caucasian | 5
  Other, Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 8
Weight [Mean (Standard Deviation); unit: lbs] | 166.8 (33.3)
Ambulatory Status [Count of Participants; unit: Participants]
  Fully Ambulatory | 3
  Partially Ambulatory | 2
  Non-Ambulatory | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device Related Serious Adverse Events
Description: Rate of participants treated with the Connected Catheter reported with a serious device related adverse event
Time Frame: 0 - 49 days
Population: This is based on the number of patients who had catheter insertion attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Connected Catheter Users
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Number of Participants With UTI (Occurrence Rate)
Description: Rate of participants treated with the Connected Catheter reported with a symptomatic urinary tract infection
Time Frame: 0 - 49 days
Population: This is based on the number of patients who had catheter insertion attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Connected Catheter Users
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Number of Participants With Lower Urinary Tract Injury
Description: Rate of participants treated with the Connected Catheter that experience a lower urinary tract injury
Time Frame: 0 - 40 days
Population: This is based on the number of patients who had catheter insertion attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Connected Catheter Users
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: From initial catheter insertion through study completion, which was up to 7 weeks.
Description: There are no significant differences in the definitions and requirements for adverse event reporting.
Arm/Group | Connected Catheter Users
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
single arm, small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04059159/Prot_SAP_000.pdf